CLINICAL TRIAL: NCT02020772
Title: Coordination Between General Practitioners and Physical Therapists in Primary Health Care for Musculoskeletal Pain: Effect on Sick Leave and Referral to Specialist Care.
Brief Title: Coordinating Teams in Primary Health Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012/1232
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Diseases
Keywords: primary health care; Physical Therapy Specialty; General Practitioners; General Practice
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- coordinating primary health care 1 (Experimental): musculoskeletal pain care by a coordinating team of one general practitioner and two physical therapists
  Interventions: Other: coordinating primary health care
- usual primary health care 1 (Active Comparator): usual care of musculoskeletal pain in general practice
  Interventions: Other: usual primary health care
- coordinating primary health care 2 (Experimental): musculoskeletal pain care by a coordinating team of one general practitioner and two physical therapists
  Interventions: Other: coordinating primary health care
- usual primary health care 2 (Active Comparator): usual care of musculoskeletal pain in general practice
  Interventions: Other: usual primary health care

INTERVENTIONS:
Other: coordinating primary health care
  Arms: coordinating primary health care 1; coordinating primary health care 2
Other: usual primary health care
  Arms: usual primary health care 1; usual primary health care 2

SUMMARY:
Patients who suffer from musculoskeletal pain often have more than one diagnosis. These patients mostly have to wait a long time for the doctor's examination and treatment, and they also often have a sick leave for a long period of time. The investigators expect that treatment and follow-up by an coordinating interdisciplinary team can improve these patients opportunity to function, increase their quality of life, and decrease their pain. The purpose of this study is to investigate if use of a coordinating interdisciplinary team in primary health care will result in reduced sick leave compared with practice as usual, and give fewer referrals to specialized health services and private rehabilitation centers. Research data will be obtained from the patients journals, questionnaires, and clinical examinations..

ELIGIBILITY:
Inclusion Criteria:

* patient in one of the participating general practices
* musculoskeletal complaints in 3 years before start of this study
* informed consent

Exclusion Criteria:

-

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 969 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
change in sick leave | 3 years
  average number of days sick leave during 3 years pre-intervention and during the first, second and third year of the study
referrals to specialist care | 3 years
  number of referrals to specialist care including private rehabilitation centers

CONTACTS AND LOCATIONS:
Overall Officials: Siv Mørkved, prof phd, Study Director — Norwegian University of Science and Technology
Locations (4):
- Norway (4):
  - Stjørdal Legesenter, Stjørdal
  - Persaunet Legesenter, Trondheim
  - Rosten Legesenter, Trondheim
  - Sjøsiden Legesenter, Trondheim

REFERENCES:
- [Result] Garnaes KK, Morkved S, Salvesen O, Tonne T, Furan L, Gronhaug G, Vasseljen O, Johannessen HH. What factors are associated with health-related quality of life among patients with chronic musculoskeletal pain? A cross-sectional study in primary health care. BMC Musculoskelet Disord. 2021 Jan 22;22(1):102. doi: 10.1186/s12891-020-03914-x. PMID 33482782
- [Derived] Garnaes KK, Morkved S, Tonne T, Furan L, Vasseljen O, Johannessen HH. Mental health among patients with chronic musculoskeletal pain and its relation to number of pain sites and pain intensity, a cross-sectional study among primary health care patients. BMC Musculoskelet Disord. 2022 Dec 22;23(1):1115. doi: 10.1186/s12891-022-06051-9. PMID 36544130